CLINICAL TRIAL: NCT05862480
Title: Use of a Hypochlorous Acid Spray Solution in the Treatment of COVID-19 Patients : COVICONTROL Study .
Acronym: COVICONTROL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, Pr Semir Nouira , Head of Emergency department , Fattouma Bourguiba Hospital, University of Monastir
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Monastir URG
Record Dates: First submitted 2023-05-12; First posted 2023-05-17 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: SARS CoV 2 Infection
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypochlorous Acid Group (HClO) (Active Comparator): Patients received one nasal spray in each nasal nostril/3 hours and two oral sprays/3 hours by a solution of hypochlorous acid (NEED DEFENDER) for 5 days
  Interventions: Other: Spray with Placebo Group
- Placebo Group (Placebo Comparator): Patients received one nasal spray in each nasal nostril/3 hours and two oral sprays/3 hours by a Placebo for 5 days .
  Interventions: Other: Spray with Hypochlorous Acid Group

INTERVENTIONS:
Other: Spray with Hypochlorous Acid Group — For Each Patient included . A prescription of a nasal spray in each nostril/3 hours and two oral sprays/3 hours by a solution of hypochlorous acid (NEED DEFENDER) for 5 days
  Arms: Placebo Group
Other: Spray with Placebo Group — For Each Patient included , A prescription of an identical to the intervention nasal spray in each nostril/3 hours and two oral sprays/3 hours by Placebo for 5 days.
  Arms: Hypochlorous Acid Group (HClO)

SUMMARY:
The objective is To evaluate the efficacy and safety of nasal spray and mouth spray application with hypochlorous acid-containing solution versus placebo as a curative treatment for hospitalized SARS-CoV-2 positive patients And for symptomatic SARS-CoV-2 positive patients followed as outpatients

DETAILED DESCRIPTION:
The COVICONTROL study is a prospective, multicenter study . It is a randomized, controlled, double-blind study.

The COVICONTROL study will be conducted in Tunisia at the COVID patient management centers in the emergency departments of Monastir (Fattouma Bourguiba) and Sousse (Hospital Of Sahloul).

After initial medical evaluation, every patient who meet the inclusion criteria, will receive randomly either A spray of solution containing hypochlorous acid or Placebo as detailed above according to the predetermined randomization.

For each patient included, one nasal spray in each nasal nostril /3 hours and two oral sprays/3 hours either by a solution of hypochlorous acid (NEED DEFENDER) or by a placebo. for 5 days None of the treating physician or nurses are aware about the nature of medication receive. In both arms, patients can receive antipyretics, antibacterials, antivirals, antifungals and anti-inflammatories at the discretion of the treating physician.

* Patients follow-up :

During the study , a research member maintains contact (face-to-face if hospitalized or by telephone if ambulatory) at D2, D3, and D5 with participating patients to ensure compliance with treatment and report on disease progression: disappearance or persistence of symptoms, need for hospitalization, need for intensive care, duration of hospitalization, need for respiratory assistance (CPAP, NIV, Optiflow, VM), duration of respiratory assistance, survival or death.

At day 3 :a nasopharyngeal swab will be taken to check the viral load using quantitative RT PCR.At D10 and D30, data on disease progression will be collected one last time.

ELIGIBILITY:
* Inclusion Criteria :

  * Patients with symptoms of COVID who are over 18 years of age and whose nasal swabs have been positive for SARS-CoV-2 based on RT-PCR testing less than 3 days .
  * Patients must have the ability to understand and be willing to sign a written informed consent document from the patient or legal representative.
  * The patient must be able and willing to comply with the requirements of this study protocol.
* Exclusion Criteria:

  1. History of allergy to hypochlorous acid solution .
  2. Oral lesions contraindicating the use of hypochlorous acid solution.
  3. Patients receiving any other investigational agent in a clinical trial.
  4. Intubated patient on mechanical ventilation or with uncontrolled disease : congestive heart failure, IDM, uncontrolled epilepsy or psychiatric illness.
  5. Uncertain patient follow-up during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
the change in viral load | 3 days
  The primary endpoint in all included patients (outpatients and inpatients ) is the change in viral load between Day 1 and Day 3

SECONDARY OUTCOMES:
Duration of symptoms | 30 days
  Evolution of symptoms : duration of symptoms , appearance and disappearance of symptoms .
Hospitalization Need for hospitalization. | 30 days
  Need for hospitalization and length of hospitalization
Need for intensive care. | 30 days
  Need for ICU
Need for ventilatory support | 30 days
  (CPAP, NIV, Optiflow, MV), and duration of ventilatory support
Contamination | 30 days
  For ambulatory patients, the secondary endpoint also includes the percentage of surrounding contamination considered on the basis of the clinic and biological confirmation if necessary.
Death | 30 days
  Death

CONTACTS AND LOCATIONS:
Overall Officials: Semir Nouira, MD, Principal Investigator — University Hospital Fattouma Bourguiba Monastir , Emergency Department .
Locations (1):
- Semir Nouira, Monastir, Tunisia